CLINICAL TRIAL: NCT02159534
Title: Multicentric Prospective Randomised Single-blind Controlled Clinical Study Assessing the Effect and the Safety of Primebrain Sensorimotor Stimulation on Neurological Development of Preterm Infants (Born Before 32 Weeks' Gestation) or Infants Born Weighing Less Than 1500 g
Brief Title: Primebrain Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Queen Fabiola Children's University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HU15/neuro/primebrain
Record Dates: First submitted 2014-06-06; First posted 2014-06-10 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Preterm Infants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Primebrain (Experimental): ' Stimulation ' Infants group will receive Primebrain stimulation whose items were selected according to a Delphi process and discussed at the European Academy of Childhood Disability (2013).
  This sensorimotor stimulation programme is administered at home by parents (trained and monitored by a physical therapist), once a day between term-age and 6 months of corrected age.
  In addition, these infants undergo systematic monitoring for preterm and infants born with low birth weight as organized in Belgium (" INAMI convention ").
  Interventions: Other: Primebrain
- usual care (Other): Infants in the comparison group receive usual care for preterm and infants born with low birth weight as organized in Belgium (" INAMI convention ").
  Interventions: Other: Primebrain

INTERVENTIONS:
Other: Primebrain — Primebrain stimulation programme aims to facilitate the infant's self-organization of postural competences by proposing varied sensorimotor experiences in a context supporting parent-child interaction.

SUMMARY:
Background : Brain vulnerability is particularly marked in preterm neonates and has long-term consequences. Unlike lesions affecting other organs, those that affect the brain can currently not 'be repaired' by producing new cells. However, exeprience-driven brain plasticity allows the brain to reorganise its connections to compensate (at least partially) the effects of an injury.

Purpose : To evaluate the influence of Primebrain stimulation programme administred by parents until 6 months post-term on motor and neurophysiological development of infants born <32 weeks' gestation or with birth weight <1500 g.

DETAILED DESCRIPTION:
Preterm and very low birth weight infants are at risk for neurodevelopmental disorders, including cerebral palsy, sensory impairment and intellectual disability. Several early intervention approaches have been designed in the hope of optimising neurological development in this context. These programmes show high variety in the type of intervention, frequency of sessions and total duration of the intervention, as well as the duration of follow-up. Depending on studies, there is an inconstant benefit on cognitive and behavioural development in the first 2 years and preschool age. According to the most recent studies, it seems important that the intervention takes into account parental mental health, focuses on parent-child interactions and lasts sufficiently long.

This prospective randomized-controlled clinical study has been designed to evaluate the effects of an additional parent-administed programme to the usual care in this developmental risk population,.

The intervention is carried out at home by parents coached by physiotherapist from term-age to 6 months of corrected age. The monitoring and evaluation period for all infants participating in the study ends at 24 months of corrected age and includes clinical, neurodevelopmental, parental stress and neurophysiological assessments using high density electroencephalography and recording of event-related potentials at term age, 3, 6, 12 ,18 and 24 months of corrected age (ActiveTwo, BioSemi).

ELIGIBILITY:
Inclusion Criteria:

* Infants born before 32 weeks of gestation or with a birth weight less than 1500 grams

Exclusion Criteria:

* Severe congenital malformation (cerebral, cardiac or within a syndrome)
* Neurodevelopmental genetic syndrome
* Cytomegalovirus, rubella or toxoplasmosis congenital infection
* Neonatal hypothyroidism
* Peripheral neurological disorder or congenital muscular disorder
* Neurodegenerative disorder

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2014-09 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Motor development using Bayley Scales of Infant Development (BSID-III) | at 24 months of corrected age.

SECONDARY OUTCOMES:
Language and cognitive development using Bayley Scales of Infant Development (BSID-III) | at 6, 12, 18 and 24 months of corrected age
Parental Stress Index (PSI), short form | at 6, 12,18 and 24 months of corrected age.

OTHER OUTCOMES:
high-density electroencephalography recording | at age-term, 3, 6, 12,18 and 24 months of corrected age
  Exploratory outcome, evaluation of neurophysiological maturation

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Fabiola Children's University Hospital, Brussels, Belgium

REFERENCES:
- [Background] Vohr BR, Wright LL, Poole WK, McDonald SA. Neurodevelopmental outcomes of extremely low birth weight infants <32 weeks' gestation between 1993 and 1998. Pediatrics. 2005 Sep;116(3):635-43. doi: 10.1542/peds.2004-2247. PMID 16143580
- [Background] Spittle AJ, Spencer-Smith MM, Eeles AL, Lee KJ, Lorefice LE, Anderson PJ, Doyle LW. Does the Bayley-III Motor Scale at 2 years predict motor outcome at 4 years in very preterm children? Dev Med Child Neurol. 2013 May;55(5):448-52. doi: 10.1111/dmcn.12049. Epub 2012 Dec 6. PMID 23216518
- [Background] Linsell L, Malouf R, Morris J, Kurinczuk JJ, Marlow N. Prognostic Factors for Poor Cognitive Development in Children Born Very Preterm or With Very Low Birth Weight: A Systematic Review. JAMA Pediatr. 2015 Dec;169(12):1162-72. doi: 10.1001/jamapediatrics.2015.2175. PMID 26457641
- [Background] Linsell L, Malouf R, Morris J, Kurinczuk JJ, Marlow N. Prognostic factors for cerebral palsy and motor impairment in children born very preterm or very low birthweight: a systematic review. Dev Med Child Neurol. 2016 Jun;58(6):554-69. doi: 10.1111/dmcn.12972. Epub 2016 Feb 10. PMID 26862030
- [Background] Linsell L, Malouf R, Johnson S, Morris J, Kurinczuk JJ, Marlow N. Prognostic Factors for Behavioral Problems and Psychiatric Disorders in Children Born Very Preterm or Very Low Birth Weight: A Systematic Review. J Dev Behav Pediatr. 2016 Jan;37(1):88-102. doi: 10.1097/DBP.0000000000000238. PMID 26703327
- [Background] Hadders-Algra M. Early brain damage and the development of motor behavior in children: clues for therapeutic intervention? Neural Plast. 2001;8(1-2):31-49. doi: 10.1155/NP.2001.31. PMID 11530887
- [Background] Ismail FY, Fatemi A, Johnston MV. Cerebral plasticity: Windows of opportunity in the developing brain. Eur J Paediatr Neurol. 2017 Jan;21(1):23-48. doi: 10.1016/j.ejpn.2016.07.007. Epub 2016 Aug 9. PMID 27567276
- [Background] Spittle A, Orton J, Anderson PJ, Boyd R, Doyle LW. Early developmental intervention programmes provided post hospital discharge to prevent motor and cognitive impairment in preterm infants. Cochrane Database Syst Rev. 2015 Nov 24;2015(11):CD005495. doi: 10.1002/14651858.CD005495.pub4. PMID 26597166
- [Background] Musacchia G, Ortiz-Mantilla S, Realpe-Bonilla T, Roesler CP, Benasich AA. Infant Auditory Processing and Event-related Brain Oscillations. J Vis Exp. 2015 Jul 1;(101):e52420. doi: 10.3791/52420. PMID 26167670
- [Background] Friel KM, Chakrabarty S, Martin JH. Pathophysiological mechanisms of impaired limb use and repair strategies for motor systems after unilateral injury of the developing brain. Dev Med Child Neurol. 2013 Nov;55 Suppl 4:27-31. doi: 10.1111/dmcn.12303. PMID 24237276
- [Background] Engle WA; American Academy of Pediatrics Committee on Fetus and Newborn. Age terminology during the perinatal period. Pediatrics. 2004 Nov;114(5):1362-4. doi: 10.1542/peds.2004-1915. PMID 15520122
- [Derived] Pelc K, Daniel I, Wenderickx B, Dan B; Primebrain group. Multicentre prospective randomised single-blind controlled study protocol of the effect of an additional parent-administered sensorimotor stimulation on neurological development of preterm infants: Primebrain. BMJ Open. 2017 Dec 3;7(12):e018084. doi: 10.1136/bmjopen-2017-018084. PMID 29203503